CLINICAL TRIAL: NCT00903396
Title: A Pilot Phase II, Randomized, Double Blind Trial of Palonosetron Versus Placebo to Prevent Radiation Therapy Induced Nausea and Vomiting
Brief Title: Palonosetron Hydrochloride in Preventing Nausea and Vomiting Caused by Radiation Therapy in Patients With Primary Abdominal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N08C2; NCI-2009-01109 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000642449 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2009-05-15; First posted 2009-05-18 (Estimated); Results first posted 2017-02-01 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-10

CONDITIONS: Anal Cancer; Carcinoma of the Appendix; Colorectal Cancer; Extrahepatic Bile Duct Cancer; Gallbladder Cancer; Gastric Cancer; Gastrointestinal Carcinoid Tumor; Liver Cancer; Nausea and Vomiting; Pancreatic Cancer; Primary Peritoneal Cavity Cancer; Small Intestine Cancer
Keywords: nausea and vomiting; gastrointestinal carcinoid tumor; anal cancer; carcinoma of the appendix; colon cancer; rectal cancer; extrahepatic bile duct cancer; gallbladder cancer; gastric cancer; liver and intrahepatic biliary tract cancer; pancreatic cancer; small intestine cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Anus Neoplasms; Appendiceal Neoplasms; Colorectal Neoplasms; Bile Duct Neoplasms; Gallbladder Neoplasms; Stomach Neoplasms; Liver Neoplasms; Nausea; Vomiting; Pancreatic Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Carcinoma, Hepatocellular | interventions — Palonosetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm I (Experimental): Patients receive palonosetron hydrochloride IV on day 1.
  Interventions: Drug: palonosetron hydrochloride
- Arm II (Experimental): Patients receive palonosetron hydrochloride IV on days 1 and 4.
  Interventions: Drug: palonosetron hydrochloride
- Arm III (Placebo Comparator): Patients receive placebo IV on day 1.
  Interventions: Other: placebo
- Arm IV (Placebo Comparator): Patients receive placebo IV on days 1 and 4.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: palonosetron hydrochloride — Given IV
  Arms: Arm I; Arm II
Other: placebo — Given IV
  Arms: Arm III; Arm IV

SUMMARY:
RATIONALE: Palonosetron hydrochloride may prevent nausea and vomiting caused by radiation therapy. It is not yet known whether palonosetron hydrochloride is more effective than a placebo in preventing nausea and vomiting.

PURPOSE: This randomized phase II trial is studying the side effects of palonosetron hydrochloride and to see how well it works in preventing nausea and vomiting caused by radiation therapy in patients with primary abdominal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the rate of complete responses, defined as no vomiting and no nausea, in patients with primary gastrointestinal and/or retroperitoneal sarcomas treated with two different dosing schedules of palonosetron hydrochloride during abdominal radiotherapy as part of their cancer treatment.
* Determine the tolerability of palonosetron hydrochloride vs placebo in these patients.
* Validate patient diaries for assessing nausea and vomiting by comparing with alternative methods for measuring nausea and vomiting in order to determine the optimal approach for future studies.

OUTLINE: Patients are stratified according to planned radiotherapy duration (< 5 weeks vs ≥ 5 weeks), planned concurrent fluorouracil ( yes vs no), and gender. Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients receive palonosetron hydrochloride IV on day 1.
* Arm II: Patients receive palonosetron hydrochloride IV on days 1 and 4.
* Arm III: Patients receive placebo IV on day 1.
* Arm IV: Patients receive placebo IV on days 1 and 4. In all arms, courses repeat weekly during radiotherapy in the absence of disease progression or unacceptable toxicity.

Patients complete nausea and vomiting questionnaires and diaries at baseline and daily during radiotherapy. Patients also complete symptom experience diaries weekly during radiotherapy.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of primary gastrointestinal and/or retroperitoneal sarcoma
* Scheduled to undergo ≥ 3000 cGy or ≥ 3 weeks of external beam radiation to the abdomen

  * Radiotherapy fields to extend between T11 and L3, and of a size ≥ 100 cm^2
* No brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Negative pregnancy test
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Able to complete questionnaire(s) alone or with assistance
* Willing to return to NCCTG enrolling institution for follow-up
* Able to reliably take oral medication (for purposes of rescue medication)
* No hypersensitivity to palonosetron hydrochloride or other selective 5-HT3 receptor antagonists
* No comorbid systemic illness or other severe concurrent disease that, in the judgment of the investigator, would make the patient inappropriate for study entry or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* No nausea ≤ 48 hours prior to study enrollment
* No history of dystonic reactions to prochlorperazine or haloperidol or related agents

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 7 days since prior agents known to have significant effects on emesis, including the following:

  * Ondansetron
  * Sedating antihistamines
  * Antipsychotics
  * Cannabinoids
  * Corticosteroids
  * Metoclopramide
  * Narcotic analgesics
  * Benzodiazepines
* More than 7 days since prior chemotherapy other than fluorouracil or capecitabine used as a radiosensitizer
* More than 7 days since of prior cetuximab
* More than 7 days since prior and no concurrent oral steroids
* No prior palonosetron hydrochloride

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2011-01 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Yvette Halyard, MD, Study Chair — Mayo Clinic
Locations (69):
- United States (69):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - Bettendorf, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Wesley Medical Center, Wichita, Kansas
  - Michiana Hematology Oncology PC - Niles, Niles, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fergus Falls Medical Group, PA, Fergus Falls, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Door County Cancer Center at Door County Memorial Hospital, Sturgeon Bay, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I | Arm II | Arm III | Arm IV
Started | 2 | 1 | 3 | 1
Completed | 2 | 1 | 3 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Not enough patients were accrued. In order to avoid identification of patients, no results will be entered.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Arm III | Arm IV | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
Age, Continuous
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (no Episodes of Nausea or Vomiting)
Time Frame: Up to 2 years
Population: Not enough patients were accrued. In order to avoid identification of patients, no results will be entered.
Arm/Group | Arm I | Arm II | Arm III | Arm IV
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Time to Treatment Failure, Defined as a Single Episode of Vomiting, Daily Nausea Score of Moderate or Greater, or Taking ≥ 3 Prochlorperazine or Haloperidol Tablets Per Day
Time Frame: Up to 2 years
Population: Not enough patients were accrued. In order to avoid identification of patients, no results will be entered.
Arm/Group | Arm I | Arm II | Arm III | Arm IV
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Proportion of Patients Reporting Treatment Failure
Time Frame: Up to 2 years
Population: Not enough patients were accrued. In order to avoid identification of patients, no results will be entered.
Arm/Group | Arm I | Arm II | Arm III | Arm IV
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Tolerability and Adverse Events as Assessed by NCI CTC v 3.0
Time Frame: Up to 2 years
Population: Not enough patients were accrued. In order to avoid identification of patients, no results will be entered.
Arm/Group | Arm I | Arm II | Arm III | Arm IV
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Average Level of Nausea Reported and the Proportion of Patients Experiencing a Complete Response Independent of Treatment Arm
Time Frame: Up to 2 years
Population: Not enough patients were accrued. In order to avoid identification of patients, no results will be entered.
Arm/Group | Arm I | Arm II | Arm III | Arm IV
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: Not enough patients were accrued. In order to avoid identification of patients, no results will be entered.
Arm/Group | Arm I | Arm II | Arm III | Arm IV
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes